CLINICAL TRIAL: NCT05521984
Title: Targeting Pediatric Brain Tumors and Relapsed/Refractory Solid Tumors With Sodium Glucose Cotransporter 2 Inhibitors (SGLT2i)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Children's Discovery Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202210013
Record Dates: First submitted 2022-08-26; First posted 2022-08-30 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Brain Tumor; Pediatric Solid Tumor
MeSH Terms: interventions — dapagliflozin; Carmustine; Topotecan; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Brain Cancer: Dapagliflozin + Standard of Care Chemotherapy (Ages 6-10) (Experimental): * Dapagliflozin will be initiated by mouth once daily at the same time as standard of care chemotherapy (carmustine).
  * Dapagliflozin 5 mg by mouth once daily on days 1-84 (duration of study)
  * All patients will stop taking dapagliflozin after 12 weeks of treatment.
  Interventions: Drug: Dapagliflozin; Drug: Carmustine
- Brain Cancer: Dapagliflozin + Standard of Care Chemotherapy (Ages 11-21) (Experimental): * Dapagliflozin will be initiated by mouth once daily at the same time as standard of care chemotherapy (carmustine).
  * Dapagliflozin will be initiated at 5 mg by mouth once daily, days 1-4 (2 weeks)
  * Dapagliflozin will be escalated to 10 mg by mouth once daily for the remaining 10 weeks (after consultation with study endocrinologist)
  * All patients will stop taking dapagliflozin after 12 weeks of treatment.
  Interventions: Drug: Dapagliflozin; Drug: Carmustine
- Solid Tumor Cancer: Dapagliflozin + Standard of Care Chemotherapy (Ages 6-10) (Experimental): * Dapagliflozin will be initiated by mouth once daily at the same time as standard of care chemotherapy (topotecan + cyclophosphamide).
  * Dapagliflozin 5 mg by mouth once daily on days 1-84 (duration of study)
  * All patients will stop taking dapagliflozin after 12 weeks of treatment.
  * Each cycle is 21 days.
  Interventions: Drug: Dapagliflozin; Drug: Topotecan; Drug: Cyclophosphamide
- Solid Tumor Cancer: Dapagliflozin + Standard of Care Chemotherapy (Ages 11-21) (Experimental): * Dapagliflozin will be initiated by mouth once daily at the same time as standard of care chemotherapy (topotecan + cyclophosphamide).
  * Dapagliflozin will be initiated at 5 mg by mouth once daily, days 1-4 (2 weeks)
  * Dapagliflozin will be escalated to 10 mg by mouth once daily for the remaining 10 weeks (after consultation with study endocrinologist)
  * All patients will stop taking dapagliflozin after 12 weeks of treatment.
  * Each cycle is 21 days.
  Interventions: Drug: Dapagliflozin; Drug: Topotecan; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Dapagliflozin — Commercially available
Drug: Carmustine — Standard of care
  Arms: Brain Cancer: Dapagliflozin + Standard of Care Chemotherapy (Ages 11-21); Brain Cancer: Dapagliflozin + Standard of Care Chemotherapy (Ages 6-10)
Drug: Topotecan — Standard of care
  Arms: Solid Tumor Cancer: Dapagliflozin + Standard of Care Chemotherapy (Ages 11-21); Solid Tumor Cancer: Dapagliflozin + Standard of Care Chemotherapy (Ages 6-10)
Drug: Cyclophosphamide — Standard of care
  Arms: Solid Tumor Cancer: Dapagliflozin + Standard of Care Chemotherapy (Ages 11-21); Solid Tumor Cancer: Dapagliflozin + Standard of Care Chemotherapy (Ages 6-10)

SUMMARY:
This is a pilot phase Ib study of the safety of dapagliflozin (in addition to standard of care treatment) for the treatment of pediatric patients with recurrent brain tumors and relapsed/refractory solid tumors. The primary hypothesis is that dapagliflozin is well-tolerated and safe to use in this patient population. The investigators also hypothesize that dapagliflozin will be efficacious as an adjunct to front-line chemotherapy assessed by decreased tumor markers mediated by its pleiotropic metabolic effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a recurrent primary brain tumor with no curative therapy available OR diagnosis of relapsed/refractory solid tumor with no curative option and has trialed past a second line of therapy.
* Measurable disease per the following:

  * For patients with brain tumors: measurable disease pediatric Response Assessment in Neuro-Oncology Criteria (RANO) criteria
  * For patients with solid tumors: measurable disease using response evaluation criteria in solid tumors (RECIST 1.1). Includes patients with diagnoses of relapsed or refractory sarcomas, neuroblastoma, and Wilms tumor. Other rare solid tumors can be discussed with study chair.
* Life expectancy > 12 weeks.
* Prior treatment with radiation alone, chemotherapy alone or combined radiation and chemotherapy is allowed.
* Patient is between 6 and 21 years old (inclusive)
* Patient is capable of swallowing whole pills
* Normal bone marrow and organ function as defined below:

  * Leukocytes ≥ 3,000/mcL
  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine ≤ IULN OR creatinine clearance ≥ 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
  * Normal room air oxygenation must be documented. If room air oxygen saturation is less than 97%, a diffusion capacity of carbon monoxide (DLCO) of greater than 80%, must be demonstrated.
* Karnofsky or Lansky performance score of ≥ 60
* Patients of childbearing potential and their partners must agree to use two forms of acceptable contraception (including one barrier method) prior to study entry and for the duration of study participation. Should a female patient or partner of a male patient become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants. All patients and/or their parents or legal guardians must sign an IRB approved written informed consent document.

Exclusion Criteria:

* Current or previous treatment with SGLT2i or thiazolidinedione.
* Current use of high dose dexamethasone (exceeding 4 mg/day). Seven days prior to start of dapagliflozin, patients receiving dexamethasone must be on a stable or decreasing dose (≤ 0.1 mg/kg/day or maximum 4 mg/day). Note that it is preferred that patients not be on dexamethasone during the study.
* A history of other malignancy with the exceptions of malignancies for which all treatment was completed at least 2 years before registration with no evidence of disease and locally treated skin squamous or basal cell carcinoma.
* Type 1 diabetes or current insulin treatment.
* History of stroke or transient ischemic attack (in the last 5 years).
* HbA1c > 8.5%. The rationale is that this is the level that would require addition of insulin. However, insulin use is excluded in this study due to the increased risk of ketoacidosis.
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to dapagliflozin or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, peripheral arterial disease, ketoacidosis, severe kidney disease (estimated glomerular filtration rate eGFR < 30 mL/min/1.73m^2), symptomatic hypotension, and chronic/frequent urinary tract infections or yeast infections.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days prior to first dose of dapagliflozin.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Number and type of adverse events experienced by participants | From start of treatment through 30 days after last day of dapagliflozin treatment (estimated to be 4 months)
  -Adverse events will be graded by CTCAE (version 5.0).

SECONDARY OUTCOMES:
Change in blood glucose | From baseline through end of treatment (estimated to be 3 months)
Change in ketones | From baseline through end of treatment (estimated to be 3 months)
Change in HbA1c | From baseline through end of treatment (estimated to be 3 months)
Changes in fructosamine | From baseline through end of treatment (estimated to be 3 months)
Changes in c-peptide | From baseline through end of treatment (estimated to be 3 months)
Changes in glucagon | From baseline through end of treatment (estimated to be 3 months)
Imaging-guided tumor response assessment | From pre-therapy to post-12 weeks of therapy
  * Tumor response will be evaluated using the updated response assessment criteria for high-grade gliomas: Response Assessment in Neuro-Oncology (RANO) working group guideline for brain tumor patients.
  * Tumor response will be evaluated using RECIST 1.1 for solid tumor patients.
Tumor response rate as measured by number of participants with complete response or partial response | From pre-therapy to post-12 weeks of therapy
  * Tumor response will be evaluated using the updated response assessment criteria for high-grade gliomas: Response Assessment in Neuro-Oncology (RANO) working group guideline for brain tumor patients.
  * Tumor response will be evaluated using RECIST 1.1 for solid tumor patients.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Cluster, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/St. Louis Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu